CLINICAL TRIAL: NCT05505214
Title: Topical Corticosteroid and Bacterial Decolonization to Prevent Radiation Dermatitis: A Randomized Controlled Trial and Quality of Life Assessment
Brief Title: Topical Steroids & Bacterial Decolonization for Radiation Dermatitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study planned but never formally submitted to the IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-14221
Record Dates: First submitted 2022-07-22; First posted 2022-08-17 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: Prior to recruitment, the study statistician conducted randomization in a 1:1:1 model, which will divide patients into three arms: (a) bacterial decolonization regimen (b) topical corticosteroid use daily or (c) topical corticosteroid use daily with antibacterial decolonization regimen.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bacterial decolonization (Experimental): Validated decolonization regimen
  Interventions: Drug: Bacterial decolonization
- Topical corticosteroid (Experimental): Mometasone furoate 0.1% cream
  Interventions: Drug: Mometasone furoate 0.1% cream
- Combination (Experimental): Validated decolonization regimen and mometasone furoate 0.1% cream
  Interventions: Drug: Bacterial decolonization and Mometasone furoate 0.1% cream

INTERVENTIONS:
Drug: Bacterial decolonization — Validated decolonization regimen consisting of intranasal 2% mupirocin ointment applied twice daily as well as chlorhexidine wash used daily to the body. This regimen is conducted by the patient for 5 consecutive days prior to the start of RT and is repeated for an additional five days every other week continuing until either the development of moist desquamation or 2 weeks after the completion of RT.
  Arms: Bacterial decolonization
Drug: Mometasone furoate 0.1% cream — Mometasone furoate 0.1% cream to be applied twice a day to the irradiated area, starting on the first day of RT and continuing until either the development of moist desquamation or 2 weeks after the completion of RT
  Arms: Topical corticosteroid
Drug: Bacterial decolonization and Mometasone furoate 0.1% cream — Validated decolonization regimen consisting of intranasal 2% mupirocin ointment applied twice daily as well as chlorhexidine wash used daily to the body. This regimen is conducted by the patient for 5 consecutive days prior to the start of RT and is repeated for an additional five days every other week continuing until either the development of moist desquamation or 2 weeks after the completion of RT. Also, mometasone furoate 0.1% cream will be applied twice a day to the irradiated area, starting on the first day of RT and continuing until either the development of moist desquamation or 2 weeks after the completion of RT
  Arms: Combination

SUMMARY:
The purpose of this study is to determine whether bacterial decolonization of the nares and skin, topical steroid therapy, or a combination of the two regimens prior to treatment with radiotherapy (RT) for breast and head and neck cancer patients can prevent grade 2 or higher grade radiation dermatitis (RD) graded via the Common Terminology Criteria for Adverse Events (CTCAE) scale and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Diagnosis of a breast or head and neck cancer with plans for fractionated RT (greater than or equal to 15 fractions in 40 Gy (Gray)) with curative intent, including post-operative patients deemed eligible for RT by their surgeons and radiation oncologists

Exclusion Criteria:

* Prior RT to the region of interest
* Existing dermatologic condition affecting the treatment area (eg: atopic dermatitis, psoriasis, and non-healing wounds; known allergy to intervention therapies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade >2 RD | At study screening/enrollment, before RT treatment has started
  Assessed via the CTCAE scale before and after RT treatment via clinical photographs graded by a blinded dermatologist (minimum grade 0, maximum grade 5, higher score is worse outcome)
Incidence of grade >2 RD | At last RT treatment session, an average of 5 weeks after treatment initiation
  Assessed via the CTCAE scale before and after RT treatment via clinical photographs graded by a blinded dermatologist (minimum grade 0, maximum grade 5, higher score is worse outcome)
Incidence of grade >2 RD | Two weeks after RT treatment completed
  Assessed via the CTCAE scale before and after RT treatment via clinical photographs graded by a blinded dermatologist (minimum grade 0, maximum grade 5, higher score is worse outcome)

SECONDARY OUTCOMES:
Quality of life Score Change | At study screening/enrollment, before RT treatment has started
  Assessed by the Skindex-16 survey given to the patient before and after RT treatment (minimum score 0, maximum score 96, higher score is worse outcome)
Quality of life Score Change | At last RT treatment session, an average of 5 weeks after treatment initiation
  Assessed by the Skindex-16 survey given to the patient before and after RT treatment (minimum score 0, maximum score 96, higher score is worse outcome)
Quality of life Score Change | Two weeks after RT treatment completed
  Assessed by the Skindex-16 survey given to the patient before and after RT treatment (minimum score 0, maximum score 96, higher score is worse outcome)

OTHER OUTCOMES:
Changes in the cutaneous microbiome and transcriptome | through study completion, an average of 2 years
  Assessed through laboratory analysis of changes in microbial skin cultures and tape-strip gene expression analysis on skin samples before and after RT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yana Kost, Study Director — Montefiore Medical Center; Lindsay Pattison, Study Director — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center-Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No